CLINICAL TRIAL: NCT00679796
Title: The Effectiveness of Varicella Vaccination in Children in Germany
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 109737
Record Dates: First submitted 2008-05-13; First posted 2008-05-19 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Varicella (Chickenpox); Chickenpox Vaccines
Keywords: varicella; case-control
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples from skin lesions
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Subjects with PCR confirmed varicella
  Interventions: Procedure: Varicella (chickenpox) lesion sampling
- Group B: Age- and practice-matched control subjects
  Interventions: Procedure: Varicella (chickenpox) lesion sampling

INTERVENTIONS:
Procedure: Varicella (chickenpox) lesion sampling

SUMMARY:
This study is undertaken to evaluate the effectiveness of currently licensed varicella vaccines under conditions of routine use in a setting where varicella vaccine is included in the childhood immunization calendar.

DETAILED DESCRIPTION:
Observational, multicenter, population-based, matched case-control study conducted in selected pediatric practices in the Munich area.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child at least one year of age, born on or after July 1 2003.
* Residence in Germany
* At least one previous well-child visit to the practice
* Written informed consent obtained from parents/guardians of the subject as per local requirements.
* Specific inclusion criterion for cases:
* Suspected primary varicella disease (i.e. chickenpox) at the time of study entry

Exclusion Criteria:

* Ineligible for varicella vaccination, due to any medical contraindication. These contraindications are:

  * History of hypersensitivity to any of the components of the vaccines
  * Congenital or acquired immunodeficiency
  * Treatment with immunosuppressive therapy
  * HIV-infected patients, when CD4 < 25% of total lymphocytes
  * Previous history of chickenpox by physician record or parental report.
  * Lack of documented vaccination history (written or computerised practice records or child's vaccination card/booklet).

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All children 12 months of age or older and born on or after 1 July 2003 whose parents contact the pediatrician at the selected sites for suspected varicella after study start. Pediatric practices in Munich and the Munich area will be initially selected.
Sampling Method: Probability Sample
Enrollment: 1012 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of PCR-confirmed varicella cases in children administered one dose of Varilrix™ (≥ 28 days after receipt of vaccine) or in unvaccinated children.

SECONDARY OUTCOMES:
Occurrence of PCR-confirmed varicella cases in children administered one dose of commercially-available varicella vaccine (≥ 28 days after receipt of vaccine) or in unvaccinated children
Occurrence of PCR-confirmed severe varicella cases in children administered one dose of Varilrix™ (≥ 28 days after receipt of vaccine) or in unvaccinated children
Occurrence of PCR-confirmed severe varicella cases in children administered one dose of commercially-available varicella vaccine (≥ 28 days after receipt of vaccine) or in unvaccinated children
Occurrence of clinical varicella cases in children administered one dose of commercially-available varicella vaccine (≥ 28 days after receipt of vaccine) or in unvaccinated children
Occurrence of clinical varicella cases in children administered two doses of commercially-available varicella vaccine (≥ 28 days after receipt of the second dose of vaccine) or in unvaccinated children

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Germany (12):
  - GSK Investigational Site, Baldham, Bavaria
  - GSK Investigational Site, Deisenhofen, Bavaria
  - GSK Investigational Site, Freising, Bavaria
  - GSK Investigational Site, Fürstenfeldbruck, Bavaria
  - GSK Investigational Site, Gilching, Bavaria
  - GSK Investigational Site, Grafing, Bavaria
  - GSK Investigational Site, Grafrath, Bavaria
  - GSK Investigational Site, Kirchheim, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Taufkirchen, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria

REFERENCES:
- [Background] Liese J et al. Effectiveness of one dose of varicella vaccine after introduction of routine varicella vaccination in Germany. Abstract presented at the 20th Congress of German Society for pediatric infectious diseases (GSPID). e.V.Mannheim, Germany, 19-21 April 2012.
- [Background] Liese J et al. Pediatric practice-based case-control study to evaluate the effectiveness of vaccination against laboratory-confirmed varicella in young children in Germany. Abstract presented at the 30th Annual Meeting of the European Society for Pediatric Infectious Diseases (ESPID) meeting, Thessaloniki, Greece 8-12 May 2012.
- [Derived] Liese JG, Cohen C, Rack A, Pirzer K, Eber S, Blum M, Greenberg M, Streng A. The effectiveness of varicella vaccination in children in Germany: a case-control study. Pediatr Infect Dis J. 2013 Sep;32(9):998-1004. doi: 10.1097/INF.0b013e31829ae263. PMID 23694831